CLINICAL TRIAL: NCT01999959
Title: Effect of Pertubation on Pregnancy Rates Before Intrauterine Insemination Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Funda Korkmaz, Dr, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3061750
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Infertility; Pertubation; Insemination
Keywords: Unexplained Infertility, Pertubation, Gonadotrophin, Ovulation Induction, Intrauterine Insemination
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pertubation performed (Experimental): Study group had pertubation and insemination
  Interventions: Procedure: Pertubation
- Pertubation not performed (No Intervention): Study group had insemination only

INTERVENTIONS:
Procedure: Pertubation — a lavage procedure of the intrauterine cavity and bilateral fallopian tubes
  Arms: Pertubation performed

SUMMARY:
To demonstrate a possible beneficial impact of pertubation we designed a randomized prospective study, in which uterine washing was administered prior to insemination in patients diagnosed with unexplained infertility.

ELIGIBILITY:
Inclusion Criteria:

* age of 18-44 years; presence of regular menstrual cycles and ovulation; absence of tubal occlusion on HSG; sperm concentration >15 million spermatozoa/ml and total sperm number >39 million/ml according to WHO criteria

Exclusion Criteria:

* the presence of endocrinologic disease; use of nonsteroidal anti-inflammatory drugs (NSAIDs) or corticosteroids; clinical findings suggestive of pelvic inflammatory disease; and the presence of undiagnosed uterine bleeding

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 6 months
  Pregnancy rate at 6 month-follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Hospital, Ankara, Cankaya, Turkey (Türkiye)

REFERENCES:
- [Derived] Yildiz F, Bozkurt N, Erdem A, Erdem M, Oktem M, Onur Karabacak R. Effect of Pertubation on Pregnancy Rates before Intrauterine Insemination Treatment in Patients with Unexplained Infertility. Int J Fertil Steril. 2014 Apr;8(1):77-84. Epub 2014 Mar 9. PMID 24695882